CLINICAL TRIAL: NCT06201767
Title: Evaluation of Abnormal Uterine Bleeding in Adolescents: A Cross Sectional Observational Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Wafaa kassem Badr, Evaluation of Abnormal Uterine Bleeding in Adolescents: A Cross Sectional Observational Study, Al-Azhar University
Other Study IDs: Evaluation of AUB
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Abnormal Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of Abnormal Uterine Bleeding in Adolescents: A Cross Sectional Observational Study

DETAILED DESCRIPTION:
Abnormal uterine bleeding (AUB) is defined as any type of bleeding in which the amount, duration, frequency and cyclicity is abnormal for a patient. It is very common symptom and it is seen in 15-20% of patient from the commencement of menarche to menopause (Singh et al., 2021). Over all prevalence of AUB varies in different population fluctuating between 10% and 30% (Sarala and Gopalan, 2020).

Although AUB may be characterized by specific menstrual abnormalities including dysmenorrhea, menorrhagia, oligomenorrhea, etc., the cause of AUB is often unknown. According to International Federation of Obstetrics and Gynecology (FIGO) the classification of AUB is based on PALMCOEIN which is an acronym for various etiologies namely polyp, adenomyosis, leiomyoma, malignancy and hyperplasia, coagulopathy, ovulatory dysfunction, endometrial disorders, iatrogenic and not otherwise classified (PALM-COEIN) (Betha et al., 2017, Sabre et al., 2021).

At the pathological level, AUB is predominantly characterized by anovulatory cycles. When ovulation does not occur, no corpus luteum is formed to produce progesterone, leading to prolonged estrogenic stimulation of the endometrium and irregular bleeding. The patient will present with polymennorrhagia, polymenorrhea and metrorrhagia (Tuchkina et al., 2020).

The non-shedding of endometrium causes an increased risk of endometrial cancer. As a clinical approach to AUB, it is essential to obtain history pertaining to puberty and menstrual history in terms of regularity, volume and duration of cycles. In addition, reproductive and sexual history plays a major role in determining the etiology of AUB in married women (Tsakiridis et al., 2022).

It is also essential to consider various non-reproductive causes of AUB, namely nutritional history, endocrine disorders, socioeconomic status and current medication history. Clinical evaluation in terms of abdominal and per vaginal examination aids in the diagnosis. But conclusive results are obtained only when the endometrium is examined either by ultrasound or histological sampling (Sabre et al., 2021, Bisht and Kalra, 2023).

Diagnosis of AUB depends upon comprehensive medical history, blood tests, imaging and histopathology. Bleeding pattern style forms the clinical basis for diagnosis of different types of AUB. Some standard menstrual index parameters are used to define bleeding pattern which are frequency, duration, regularity, volume and intermenstrual bleeding (Munro et al., 2018, Singh et al., 2019).

In majority of the patients, AUB is a recurring problem and therefore, poses a challenge to the care providers in terms of clinical management. Moreover, its consequences are increasingly incriminating on the quality of life of these reproductive women, due to the impact on general health and wellbeing (Sarala and Gopalan, 2020).

Although studies have been done on evaluating the endometrium for various pathologies, there is still a vacuum with regards to the clinical presentation and correlation of AUB (Marnach and Laughlin-Tommaso, 2019, Van Den Bosch et al., 2021, Heremans et al., 2022). Clinical correlation plays a significant role in limited resource settings, especially in developing economies like Egypt, and an in-depth evaluation of clinical presentation of AUB will aid the primary care physician to detect AUB at an early stage and appropriate referral for advanced care.

ELIGIBILITY:
Inclusion Criteria:

* - Adolescent female 10- 19 years old
* Any abnormal uterine bleeding

Exclusion Criteria:

* Adolescent female with normal uterine bleeding
* Primary amenorrhea

Ages: 10 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Detailed History tacking including:
  * Personal history age, residence, marital status, special habits, menstrual history
  * Present history
  * Obstetric history for married adolescents for gravity, parity, pregnancy complication
  * Past history and gynecological conditions as myomectomy, ovarian cystectomy
  * Family history for bleeding tendency as von willebrand disease or coagulopathies
  * Examination:
  * Investigations Laboratory like complete blood picture, coagulation profile, hormonal analysis (TSH, prolactin, LH, FSH), assessment von wollbrand disease by von wollbrand factor antigen and activity Ultrasonography for evaluation
Sampling Method: Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of abnormal uterine bleeding and determining the type of abnormality. | baseline

SECONDARY OUTCOMES:
Analysing various cause of AUB in this age according to FIGO classification system. Analysing various cause of AUB in this age according to FIGO classification system | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ali Mohamed, professor, Study Director — Al-Azhar University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Betha, K., Malavatu, L. & Talasani, S. 2017. Distribution of causes of abnormal uterine bleeding using new FIGO classification system-PALM COEIN: a rural tertiary hospital based study. International Journal of Reproduction, Contraception, Obstetrics and Gynecology, 6, 3523-3528. Bisht, D. S. & Kalra, R. 2023. Endometrial Biopsy Audit and its Clinico-Pathological Correlation in Patients with Abnormal Uterine Bleeding in a Zonal Care Centre. International Journal of Contemporary Pathology, 9. Heremans, R., Van Den Bosch, T., Valentin, L., et al. 2022. Ultrasound features of endometrial pathology in women without abnormal uterine bleeding: results from the International Endometrial Tumor Analysis study (IETA3). Ultrasound in Obstetrics & Gynecology, 60, 243-255. Marnach, M. L. & Laughlin-Tommaso, S. K. Evaluation and management of abnormal uterine bleeding. Mayo Clinic Proceedings, 2019. Elsevier, 326-335. Munro, M. G., Critchley, H. O., Fraser, I. S., et al. 2018. The two FIGO systems for normal and abnormal uterine bleeding symptoms and classification of causes of abnormal uterine bleeding in the reproductive years: 2018 revisions. International Journal of Gynecology & Obstetrics, 143, 393-408. Sabre, A., Serventi, L., Nuritdinova, D., et al. 2021. Abnormal uterine bleeding types according to the PALM-COEIN FIGO classification in a medically underserved American community. Journal of the Turkish German Gynecological Association, 22, 91. Sarala, V. & Gopalan, U. 2020. Clinical pattern and presentation of abnormal uterine bleeding. International Journal of Reproduction, Contraception, Obstetrics and Gynecology, 9, 126-129. Singh, N., Faruqi, M. & Pradeep, Y. 2019. Clinico epidemiological profile of abnormal uterine bleeding in reproductive womens: a cross sectional study. International Journal of Reproduction, Contraception, Obstetrics and Gynecology, 8, 4396. Singh, P. B., Purwar, R. & Mall, R. P. 2021. Clinical spectrum and causes of abnormal uterine bleeding in reproductive age according to two FIGO systems. The New Indian Journal of OBGYN, 8, 105-106. Tsakiridis, I., Giouleka, S., Koutsouki, G., et al. 2022. Investigation and management of abnormal uterine bleeding in reproductive-aged women: a descriptive review of national and international recommendations. The European Journal of Contraception & Reproductive Health Care, 27, 504-517. Tuchkina, I. O., Vygivska, L. A. & Novikova, A. A. 2020. Abnormal uterine bleeding in adolescents: current state of the problem. Wiadomości Lekarskie, 73, 1752-1755. Van Den Bosch, T., Verbakel, J., Valentin, L., et al. 2021. Typical ultrasound features of various endometrial pathologies described using International Endometrial Tumor Analysis (IETA) terminology in women with abnormal uterine bleeding. Ultrasound in Obstetrics & Gynecology, 57, 164-172.